CLINICAL TRIAL: NCT02620735
Title: Innovative Smart-phone-enabled Health Coaching Intervention (iMOVE) to Promote Long-term Maintenance of Physical Activity Behavior in Breast Cancer Survivors: Study Protocol for a Feasibility Pilot Randomized Controlled Trial
Brief Title: Smart-phone Health Coaching Intervention to Promote Maintenance of Exercise in Breast Cancer Survivors:Protocol
Acronym: iMOVE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Canadian Breast Cancer Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 13-6157-DE
Record Dates: First submitted 2015-11-19; First posted 2015-12-03 (Estimated); Last update posted 2019-07-08 (Actual); Status verified 2019-07

CONDITIONS: Breast Neoplasms
Keywords: Exercise, health coaching, RCT, telehealth,
MeSH Terms: conditions — Breast Neoplasms; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exercise Only (Active Comparator): Participants receive 12-weeks PA training (1x/week - 60 min) group sessions with a CEP/RKin, and a progressively structured home-based exercise program based on the American College of Sports Medicine (ACSM) guidelines.It combines aerobic-resistance exercise with flexibility training, and progresses towards increased in intensity and improved fitness. The goal is at least 150 min/week of moderate-intensity aerobic activity. Participants are also asked to complete 3-5 additional home-based sessions of aerobic, and resistance activities each week. Initial intensity is based on the performance of the exercises during a group session and is self-monitored via the 10-point rating of perceived exertion, with a prescribed training zone of 4-7.
  Interventions: Behavioral: Exercise Only
- Exercise + iMOVE (Experimental): Participants will receive the same exercise program at the Exercise Only group + 1) one-on-one telephone-based counselling (10 x 30-minute telephone: weeks 1, 2, 3, 4, 5, 6, 8, and 12 (during the exercise program) and at weeks 20,28 (post-exercise program booster sessions)); 2) supportive software on smart-phone devices (the HealthCoach program), 3) use of Fit-bit and corresponding software. The iMOVE intervention was designed to enhance sustained behavior change. The theoretical constructs employed are based on promoting motivation and establishing: a) exercise self-efficacy, b) social support for exercise and c) positive exercise-induced feelings during the acute intervention (12 weeks) and post-exercise program period (6 months).
  Interventions: Device: Fit bit Device; Behavioral: Exercise Only; Behavioral: Connected Wellness HealthCoach Software; Behavioral: Health Coaching

INTERVENTIONS:
Device: Fit bit Device — Use of the fit bit flex for the duration of the study. Measures steps and sleep. Health Coaching
  Arms: Exercise + iMOVE
Behavioral: Exercise Only — 12 week exercise program
Behavioral: Connected Wellness HealthCoach Software — Use of the app on Smart-phones and an online platform. Measures the following factors: Mood, Pain, energy,exercise not picked up by Fit bit.
  Arms: Exercise + iMOVE
Behavioral: Health Coaching — 10 over the phone health coaching sessions.
  Arms: Exercise + iMOVE

SUMMARY:
While physical activity (PA) appears to play an important role in disease control and the promotion of long-term health and well-being of cancer survivors, the large majority of breast cancer survivors are not physically active. Addressing this problem requires exercise promotion and an additional method of supporting long term exercise adherence. In response, an innovative health coaching intervention which uses mobile technology (iMOVE) to promote long-term PA in breast cancer survivors (BrCa) was developed. Project description: 107 inactive BrCa survivors will be randomized to receive a 12-week exercise program (CONTROL) OR a 12 week exercise program plus a concurrent health coaching program (iMOVE) consisting of telephone-based coaching sessions and interactive software delivered through a smart-phone and Fit-bit (wearable fitness technology) (INTERVENTION). Information on the feasibility and acceptability of the methods and intervention and examine the impact on fitness (primary), patient-reported, anthropometric, and physical (secondary) outcomes will be collected. Impact and relevance: PA has increasingly been identified as a modifiable factor that has the potential to impact cancer outcomes and improve quality of life. iMOVE is an innovative intervention with the potential to promote and maintain physical activity for breast cancer survivors. This study will be the first step in the evaluation of iMOVE and will help to determine whether a larger randomized controlled trial is needed.

DETAILED DESCRIPTION:
In order to advance PA adoption and maintenance in BrCaS, an innovative health coaching intervention which uses mobile, wearable technologies (iMOVE) was developed. This pilot study will evaluate iMOVE and inform the design of a larger pragmatic randomized controlled trial (RCT).

Main Hypotheses: 1) The study will be adequately recruit (>40%) and retain (>75%) participants, and 2) the intervention will be highly acceptable to participants and result in substantial sustained fitness improvements.

Aims of the Pilot Study Aim 1: To evaluate feasibility of the methods employed as defined by a) ability to recruit >40% of those eligible; b) adequate retention, operationalized as 6-month assessment completion by >75% of participants; c) adequate adherence, operationalized as ≥70% of intervention components completed.

Aim 2: To evaluate acceptability feedback for the final refinement and optimization of the intervention.

Aim 3: To determine preliminary intervention efficacy on fitness (primary) and on patient-reported, anthropometric and physical (secondary) outcomes.

This pilot RCT enrolls inactive BrCa survivors (BrCaS) stratified by age (<55/> 55 yr) and adjuvant hormone therapy (AHT) exposure [AHT yes/AHT no]. Recruitment is undertaken at the Princess Margaret Cancer Centre (PM) while interventions occur at the Electronic Living Library for Cancer Survivorship Research (ELLICSR), the Cancer Survivorship and Wellness Centre at the Toronto General Hospital (TGH). Both PM and TGH are members of the University Health Network in Toronto, Ontario and research ethics board approval was obtained from the University Health Network (13-6157-DE).

Patients, identified from weekly-generated clinic lists and chart reviews, are approached by a member of their clinical team and those interested meet with a research assistant who explains the study and screens for eligibility. Participants are also recruited by advertisement flyers located in common hospital areas. Eligibility is ascertained over-the-phone when possible, with written consent obtained in person prior to randomization.

After participants complete baseline questionnaires and initial physiological assessments, stratification-related data (age, AHT status, eligibility ID) is emailed to a biostatistician in the Department of Biostatistics at PM who performs randomization and sends a Study ID with experimental or control group allocation.

Intervention Participants in the experimental and control conditions receive 12-weeks of PA training that includes once weekly group sessions with a certified exercise physiologist (CEP) and a registered kinesiologist (RKin), and a progressively structured, individualized home-based exercise program. The program is based on the American College of Sports Medicine (ACSM) guidelines and modeled after a successful, theory-based, mixed-modality program developed by Santa Mina et al. The individually-tailored exercise prescription combines aerobic-resistance exercise with flexibility training, and progresses under the CEP/RKin's guidance towards increases in intensity and improved fitness. Based on ACSM guidelines the goal is at least 150 minutes per week of moderate-intensity aerobic activity. Carefully calibrated increases in exercise volume over 12 weeks is intended to minimize injury risks and potential discouragement over variations in progress. Weekly group sessions of 60 minutes duration (including aerobic and resistance training) optimize social reinforcements. Participants are provided choices of days/times for the weekly supervised sessions. Participants are also asked to complete 3-5 additional home-based sessions of aerobic (e.g. brisk walking, cycling), and resistance activities (using elastic bands and body weight lift exercises) each week. Initial intensity is based on the performance of the exercises during a group session with the CEP/RKin and is self-monitored via the 10-point rating of perceived exertion, with a prescribed training zone of 4-7. Participants keep a weekly exercise log and review it at each face-to-face meeting with the CEP/RKin. All participants are provided with an exercise manual that includes exercise descriptions with instructive photographs, exercise safety guidelines, and stretching instructions. After all participants have been recruited and enrolled, semi-structured exit interviews will be completed with N = 25 participants at week # of the intervention.

Experimental Group To promote adoption and maintenance of fitness and PA levels, experimental group participants are concurrently provided with a smart-phone-based health coaching intervention (iMOVE). iMOVE has three components: 1) one-on-one telephone-based counselling; 2) supportive software on smart-phone devices (the HealthCoach program), 3) use of Fit-bit and corresponding software. The iMOVE intervention was designed to enhance sustained behavior change re: PA, integrating several elements under the terms smart-phone-based health coaching, and is based on multiple behavior-change theories, specifically Motivational Interviewing (MI); Cognitive Behavioral Therapy (CBT), TPB, TTM ; Social Learning Theory and Relapse Prevention Therapy. Once decisions to regularly exercise are made (TTM), participants elicit support from influential individuals (TPB-SLT) and undertake sessions that progress to higher fitness levels (SLT-progressive mastery). Participants are additionally supported by observations of peer progress and peer-familial social supports when disruptions in regularity occur (SLT - social modeling/social support). The careful monitoring of subjective states sensitizes subjects to regulatory effects (elevated mood, reduced fatigue), preparing them to confront adherence disruptions with a re-decision process (TTM) and re-mobilization (RPT-TTM). Instead of reacting with self-blame, temporary setbacks become prolapses such that trial-and-error learning builds future success (RPT). Consistently adherent behaviour ultimately includes non-adherent lapses and recoveries of effective routines (TTM-RPT). The theoretical constructs employed are based on promoting motivation and establishing: a) exercise self-efficacy, b) social support for exercise and c) positive exercise-induced feelings during the acute intervention (12 weeks) and post-exercise program period (6 months).

The telephone-based health coaching portion of iMOVE includes 10 x 30-minute telephone calls with a trained health coach scheduled at weeks 1, 2, 3, 4, 5, 6, 8, and 12 (during the exercise program) and at weeks 20 and 28 (post-exercise program booster sessions). The calls focus on the assessment of motivation, promotion of self-efficacy and collaborative problem solving. Telephone based counselling provides several advantages over face-to-face counselling, notably the potential for multi-regional population access given the telephone is a widely available communication medium that requires no travel by users or providers. The focus of is on assessing motivation, promoting self-efficacy and mutual problem solving to promote PA maintenance. The selected schedule provides support while building autonomy and independent motivation. The primary approach used by the health coaches is MI and CBT. MI is a collaborative, person-centered counselling method that elicits and strengthens motivation for behaviour-change by resolving ambivalence. MI has demonstrated effectiveness in increasing PA in cancer survivors and other chronic conditions and some MI-related effects have been shown to endure for two years post-intervention. Whenever self-efficacy appears impeded by distorted cognitions, CBT principles are applied, particularly to positively affect mood fluctuations. Distorted cognitions prevent enactment of health-behaviors and can drive unhealthy behaviors. With CBT, distorted cognitions can be modified, preventing or ameliorating associated negative emotional responses. Telephone-based interventions have been effective and acceptable to BrCa patients and useful in delivering MI-type/CBT interventions, include Diabetes health coaching study. As common with MI and CBT interventions, a handbook was created, which includes global objectives per session with relevant clinical tools that health coaches use to navigate sessions. An agenda for each session is facilitated by the health coach based on patient goals, activity, and motivation as collected by the software (between-sessions) and during sessions. Health coaches with a counselling background in MI and CBT and experience working with BrCa populations, receive clinical supervision by a Registered Psychologist and a Motivational Interviewing Network of Trainers (MINT) certified trainer. Fidelity of the intervention is assessed by routine review of implementation fidelity.

In addition to the scheduled telephone-based sessions, participants interact with the HealthCoach software via smart-phone. This software, previously successfully tested with participants diagnosed with type II diabetes, is tailored for BrCa. It provides participants with specific health tips (delivered by video and verbally), and the ability to track PA, nutrition, pain and psychological well being (mood, energy); it also supports goal setting (with selective automatic daily/hourly reminders). All entries into the software are time-stamped, allowing for graph creation over time which combines multiple trackers, enabling participants and health coaches to see how health indicators change in relation to active health practices. The use of the software's capabilities of initiating contact with the health coach via text messaging will be quantified and recorded. When a patient texts their health coach via the app the health coach records the number of times contacts takes place and text message content. Confirmation of the text message will be provided but will direct the patient to discuss the matter further during the next phone session. Any content that indicates a medical or emergency need will be dealt with immediately and contact with the patient will be made.

The use of the Fit-bit flex provides another way to help participants remain adherent to PA routines. Its real time feedback on activity (lights on device indicate % completion of the pre-set 10000 step goal), as well connectivity to the Connected Wellness platform allows the participant and the Health Coach to jointly explore how PA achieved by walking is being integrated into the participants life. It has a simple display of 5 LED lights which indicate the number of steps taken daily, and it vibrates to indicate that pre-set goals of 10000 steps have been reached. The lights also indicate battery level. The Fit-bit Flex includes a specialized universal series bus (USB) charger; with a battery charge that lasts for five to seven days, and takes one to two hours to charge. The tracker measures steps taken, and combines it with user data to calculate distance walked, calories burned, and activity duration-intensity. It also measures sleep quality by tracking periods of restlessness, how long it takes the wearer to fall asleep, and how long they are actually asleep. The Fit-bit has its own app which the user can use to monitor their own activity.

ELIGIBILITY:
Inclusion Criteria:

* Within 2 years of completion of adjuvant therapy, with the exception of hormone therapy, for early stage (0-IIIA) BrCa
* Baseline participation of < 60 min of weekly pre-planned PA
* Physician permission for moderate PA participation 4)Able to read and write English
* Able to attend in-person exercise training sessions and physiologic assessments at prescribed intervals.

Exclusion Criteria:

* Plans to join a weight-loss or exercise program within 9 months)
* Current pregnancy or planned pregnancy within 9 months)
* Planned surgery during study; 4) not willing to be randomized.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2014-12 (Actual); Primary Completion 2019-07 (Actual); Study Completion 2019-07 (Actual)

PRIMARY OUTCOMES:
Recruitment Rate | Through study completion, average of 2 years
  Based on CONSORT criteria, a screening log enables data collection on eligible consented (pre- and post-initial screen) and non-recruited participants with reasons for non-recruitment recorded.
Retention Rate | Through study completion, average of 2 years
  To optimize retention and prevent attrition, stability (with some flexibility) is aimed for with group exercise in terms of class time/location, combined with careful selection and training of Health Coaches, short referral times
Capture of Outcomes - proportion of participants from whom complete information is derived on clinical outcomes. | through study completion, average of 2 years
  As another major facet of feasibility, we assess the proportion of participants from whom complete information is derived on clinical outcomes, at which assessment time-points and then document rates of missing data. This outcome is measured in terms of frequency of completion not in the units of the measures themselves.
Treatment Implementation and Fidelity - length, number and quality of health coaching phone sessions | through study completion, average of 2 years
  For the experimental group, health coaching session lengths/numbers are recorded. The health coach will document use of health coaching techniques and tools, and the barriers identified. Use of the health coaching software is stored on the secure server and will be used to measure and analyze self-report and health coach activity.
Acceptability:Participants perceptions regarding their experience of the study and if they liked it | through study completion, average of 2 years
  To assess acceptability and inform future refinement, telephone interviews will be conducted with a purposefully selected sub-sample of experimental participants following intervention completion. The goal of the qualitative interviews is: 1) to explore participant perspectives of feasibility/acceptability of the health coaching intervention, and 2) to gain an understanding of specific experiences/attitudes among those successful and unsuccessful at PA maintenance PA. An interpretive description qualitative methodology will be used to meet this objective [154]. We will purposefully select participants, ensuring equal representation from participants who report exercise behavior has increased or decreased or stayed the same. We anticipate interviewing between 6-10 participants per group. A record of participation in the latter will be kept to distinguish these participants from those who were not chosen to participate. The semi-structured interviews will be 45-60 minutes in length.

SECONDARY OUTCOMES:
Change in Cardiorespiratory fitness - "VO2"(oxygen consumption) Peak (mlO2/kg/min) | baseline, 12 week, and 36 weeks
  assessed by a physician-supervised graded exercise test using the modified Bruce protocol[155]. Directly measured "VO2" peak (mlO2/kg/min) and anaerobic threshold (AT) is obtained using a metabolic cart ("Parvomedics Trueone 2400" - name of machine) with continuous gas exchange analysis during incremental treadmill walking to peak capacity. Subjects perform an incremental ramp test to the limit of tolerance. A ramp slope based on sex, age and physical fitness of subjects is set to facilitate a test duration of 10-15 minutes. The limit of tolerance is defined as the point at which subjects cannot maintain current speed (miles per hour) and incline (%) despite encouragement from the CEP/RKin. Blood pressure and arterial oxygen saturations are measured at rest and during exercise. Absolute and relative test termination criteria are based on standardized guidelines[156].
  Absolute and relative test termination criteria will be based on standardized guidelines
Change in exercise frequency - Leisure-Time Exercise Questionnaire (LTEQ) | baseline, 12 week, and 36 weeks
  Leisure-Time Exercise Questionnaire (LTEQ)- assesses exercise frequency and intensity;; assesses indices of state anxiety
Change in body mass index (kg/m2) | baseline, 12 week, and 36 weeks
  Body composition is assessed by body mass index (BMI). BMI is calculated using the participant's weight and height (BMI = weight [kg]/height [m]2). WC is measured with anthropometric tape according to protocols defined by the World Health Organization (tape placed horizontally mid-way between the bottom of the rib cage and the iliac crest) and body fat percentage is measured using bioelectric impedance analysis [156] . To assess musculoskeletal function, grip strength is measured with a Jamar Dynamometer using the standard protocol.
Change in waist circumference (WC) (cm) | baseline, 12 week, and 36 weeks
  Waist circumference is measured using anthropometric tape according to protocols defined by the World Health Organization (tape placed horizontally mid-way between the bottom of the rib cage and the iliac crest) and is measured in cm. and body fat percentage is measured using bioelectric impedance analysis [156] . To assess musculoskeletal function, grip strength is measured with a Jamar Dynamometer using the standard protocol.
Change in quality of life - Functional Assessment of Cancer Therapy-Breast (FACT-B) | baseline, 12 weeks, 36 weeks
  Functional Assessment of Cancer Therapy - Breast (FACT-B) - assesses quality of life
Change in indices of anxiety - Spielberger's State-Trait Anxiety Inventory-State (STAI-S) | baseline, 12 weeks, 36 weeks
  Assesses indices of state anxiety
Change in state of depressive symptoms - The Center for Epidemiological Studies-Depression Scale Short Form (CESD-SF) | baseline, 12 weeks, 36 weeks
  The Center for Epidemiological Studies-Depression Scale Short Form (CESD-SF)- measures state of depressive symptoms
Change in breast cancer related fatigue - Functional Assessment of Cancer Therapy-Fatigue (FACT-F) subscale | baseline, 12 weeks, 36 weeks
  Functional Assessment of Cancer Therapy-Fatigue (FACT-F) subscale - assesses BrCa related fatigue;
Change in breast cancer related physical symptoms - The Breast Cancer Prevention Trial (BCPT) Symptoms Scale | baseline, 12 weeks, 36 weeks
  The Breast Cancer Prevention Trial (BCPT) Symptoms Scale - measures BrCa related physical symptoms;
Change in fear of recurrence - Fear of Recurrence Questionnaire (FRQ) | baseline, 12 weeks, 36 weeks
  Fear of Recurrence Questionnaire (FRQ) - provides measures on a 5-point Likert scale concerning fear of cancer recurrence
Group cohesion measure - Physical Activity Group Environment Questionnaire (PAGEQ) | 12 weeks
  Physical Activity Group Environment Questionnaire (PAGEQ) will be used to measure group cohesion
Change in body fat percentage (%) | baseline, 12 weeks, 36 weeks
  Body fat percentage is measured using bioelectric impedance analysis(156).
Change in grip strength (kg of force) | baseline, 12 weeks, 36 weeks
  To assess musculoskeletal function, grip strength is measured with a Jamar Dynamometer using the standard protocol.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer M Jones, PhD, Principal Investigator — University Health Network, Toronto
Locations (1):
- ELLICSR, Toronto General Hospital 200 Elizabeth St., Toronto, Ontario, Canada

REFERENCES:
- [Derived] Ritvo P, Obadia M, Santa Mina D, Alibhai S, Sabiston C, Oh P, Campbell K, McCready D, Auger L, Jones JM. Smartphone-Enabled Health Coaching Intervention (iMOVE) to Promote Long-Term Maintenance of Physical Activity in Breast Cancer Survivors: Protocol for a Feasibility Pilot Randomized Controlled Trial. JMIR Res Protoc. 2017 Aug 24;6(8):e165. doi: 10.2196/resprot.6615. PMID 28838886